CLINICAL TRIAL: NCT05754684
Title: Quadruple Immunotherapy for Paediatric Patients With Relapsed or Refractory Neuroblastoma
Brief Title: Quadruple Immunotherapy for Neuroblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hong Kong Children's Hospital (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheuk Ka Leung Daniel, Consultant, Hong Kong Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HKCH-REC-2021-007
Record Dates: First submitted 2022-11-18; First posted 2023-03-06 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-03

CONDITIONS: Neuroblastoma Recurrent
MeSH Terms: interventions — dinutuximab; Interleukin-2; aldesleukin; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Spironolactone; naxitamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Quadruple immunotherapy
  Interventions: Biological: Natural killer cell; Drug: Dinutuximab beta; Drug: Interleukin-2; Drug: Granulocyte-Macrophage Colony-Stimulating Factor; Drug: Spironolactone; Drug: Naxitamab

INTERVENTIONS:
Biological: Natural killer cell — Natural killer cells isolated from HLA-haploidentical relative donor
  Other Names: NK cell
Drug: Dinutuximab beta — Dinutuximab beta iv for 5 days
  Other Names: Ch14.18
Drug: Interleukin-2 — Interleukin-2 sc alternate day for 6 doses
  Other Names: Aldesleukin
Drug: Granulocyte-Macrophage Colony-Stimulating Factor — Granulocyte-macrophage colony-stimulating factor sc daily till ANC >2,000/mm3
  Other Names: Sargramostim
Drug: Spironolactone — Spironolactone po three time daily
  Other Names: Aldactone
Drug: Naxitamab — Naxitamab iv for 4 days (as alternative for dinutuximab)
  Other Names: hu3F8

SUMMARY:
This is a single-arm clinical trial to evaluate the efficacy and safety of quadruple immunotherapy with natural killer (NK) cells, anti-GD2 antibody, cytokines (interleukin-2 (IL-2) and granulocyte-macrophage colony stimulating factor (GM-CSF)) and retinoid X receptor gamma (RXRg) agonist spironolactone for paediatric patients with relapsed or refractory neuroblastoma.

DETAILED DESCRIPTION:
Included patients will receive intravenous infusion of donor NK cells on day 0, and anti-GD2 antibody (dinutuximab) on day -6 to day -2. IL-2 will be given subcutaneously on day -1, day +1, day +3, day +5, day +7, and day +9. Subcutaneous injection of GM-CSF will be started on day 0, given daily till neutrophil count >1000/mm3. Spironolactone will be started orally on day -1, given three times daily till cessation of GM-CSF.

Alternative anti-GD2 antibody (Naxitamab) can be used instead of dinutuximab, to be given on day -5, day -3, day +1 and day +3.

ELIGIBILITY:
Inclusion Criteria:

* relapsed or refractory neuroblastoma
* Adequate organ function: creatinine clearance ≥40 ml/min/1.73m2, total bilirubin ≤3 times upper limit of normal and ALT ≤500 IU/L, left ventricular shortening fraction ≥25%, and oxygen saturation ≥92% in room air
* Karnofsky or Lansky performance status score ≥50
* Has an appropriate HLA-haploidentical NK-cell donor available

Exclusion Criteria:

* Pregnant or lactating woman
* HIV infection
* Patients for whom conventional treatment is deemed more appropriate
* Patients who are unlikely to benefit, e.g., terminal malignancy with life expectancy <1 month

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who have objective response in the tumor | 1-2 months
  Objective response = complete response + partial response + minor response + stable disease

SECONDARY OUTCOMES:
Overall survival at 1 year | up to 1 year
  From the date of treatment start until the date of death from any cause, assessed up to 1 year
Progression-free survival | up to 1 year
  From date of treatment start until the date of first documented progression or the date of death from any cause, whichever comes first, assessed up to 1 year
Proportion of patients who have tumor relapse | up to 1 year
  relapse = reappearance of tumor after complete response
Number of patients who experience adverse events | up to 1 month
  Adverse events are graded according to Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events version 5 (CTCAEv5)
Percentage of donor NK cells | up to 1 year
  Percentage of donor natural killer cells in the recipient's blood will be evaluated weekly from the date of NK cell infusion for 4 weeks, then every 2 weeks till donor NK cells are undetectable

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cheuk, Principal Investigator — Hong Kong Children's Hospital
Locations (1):
- Hong Kong Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No